CLINICAL TRIAL: NCT02089854
Title: Evaluation of Adjuvant Endocrine Therapy for Operable ER-beta Positive, ER-alpha/PR Negative, Her-2 Negative Breast Cancer Patients
Brief Title: Adjuvant Endocrine Therapy for Estrogen Receptor-beta Positive Triple Negative Breast Cancer
Acronym: AETNBC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-breast-TNBC
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Female Breast Cancer
Keywords: triple negative breast cancer; estrogen receptor-beta; endocrine therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Toremifene; Anastrozole

ARMS (2):
- endocrine therapy (Experimental): toremifene 60mg PO. per day for premenopausal and perimenopausal patients; anastrozole 1mg PO. per day for postmenopausal patients
  Interventions: Drug: Toremifene; Anastrozole
- observation (No Intervention)

INTERVENTIONS:
Drug: Toremifene; Anastrozole — Toremifene 60mg PO. per day for premenopausal and perimenopausal patients; Anastrozole 1mg PO. per day for postmenopausal patients
  Arms: endocrine therapy

SUMMARY:
The study is a prospective multi-center randomized control clinical trial which is sponsored by the researchers. The purpose of this study is to determine the effectiveness of adjuvant endocrine therapy for operable ER-beta positive, ER-alpha/PR negative, Her-2 negative breast cancer(triple negative breast cancer, TNBC) patients. The ER-beta positive TNBC patients who had undergone modified radical mastectomy or breast-conserving surgery were randomly (1:1) enrolled to receive toremifene (60 mg per day for premenopausal and perimenopausal patients) /anastrozole(1mg per day for postmenopausal patients) or observation within 4 weeks after adjuvant chemotherapy and/or radiation therapy if necessary.The follow-up time will be at least five years. The disease free survival(DFS) and overall survival(OS) between endocrine group and observation group will be compared to evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent.
* The patients present with histologically proven operable invasive breast cancers without distant metastasis.
* The breast tumor's positive ER/PR rate is <1%, and positive ER-beta rate is ≥1% by immuno-histochemistry(IHC).
* The patients have no history of neoadjuvant hormone therapy.
* The patients' Karnofsky performance score ≥70%.
* Female patient who is ≥ 18yrs, and ≤ 80yrs.
* The patients are non-pregnant, and disposed to practice contraception during the whole trial.
* The patients underwent neoadjuvant chemotherapy plus surgery or directly modified radical mastectomy or breast-conserving surgery (plus sentinel lymph node biopsy or axillary lymph node dissection) after diagnosis of breast cancer.
* The patients underwent chemotherapy, radiation therapy after surgery according to the 2013 NCCN guideline.
* The results of patients' blood tests are as follows:

Hb≥90g/L; WBC≥4.0×109/L; Neutrophils≥1.5×109/L; Plt≥100×109/L; alanine aminotransferase(ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal(ULN); total bilirubin(TBIL) ≤ 1.5×ULN; Creatinine ≤ 1.25×ULN.

Exclusion Criteria:

* The patients have a previous history of invasive malignant disease (breast cancer at any time, other malignant disorders within the past 10 years excluding squamous or basal-cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied).
* The patients have any severe concomitant disease which will place the patient at unusual risk or confound the results of the trial.
* The patients have history of neoadjuvant hormone therapy.
* The patients are undergoing current administration of anti-cancer therapies, or are attending other clinical trials.
* The patients are pregnant or lactational, or they refuse to practice contraception during the whole trial.
* The patients are unwilling to stop any hormonal drug including hormone replacement therapy(HRT).
* The patients can't understand the written informed consent; such as they have dementia.
* The patients have allergic history or contraindication of toremifene/anastrozole.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China